CLINICAL TRIAL: NCT07406399
Title: A Randomized Controlled Study of Low Concentration Atropine Combined With Soft Contact Lens in Controlling Myopia Progression in Children With High Myopia
Brief Title: Low Concentration Atropine Combined With Soft Contact Lens in Controlling Myopia Progression in Children With High Myopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Mengtian Kang, attending physician, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TREC2022-KY110
Record Dates: First submitted 2026-02-01; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: High Myopia; Low Concentration Atropine; Soft Contact Lens; Children
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Generation of random sequences, determination of random number grouping, and inclusion of subjects by different staff members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- combination therapy group (Experimental): 40 patients in combination therapy group received atropine 0.04% plus soft peripheral defocus contact lenses
  Interventions: Device: soft peripheral defocus contact lenses; Drug: Atropine 0.04%
- atropine monotherapy group (Experimental): 40 patients in atropine monotherapy group received atropine 0.04% plus spectacles
  Interventions: Drug: Atropine 0.04%; Device: Single Vision Spectacles
- control group (Placebo Comparator): 40 patients in control group received atropine 0.01% plus spectacles
  Interventions: Drug: Atropine (0.01%); Device: Single Vision Spectacles

INTERVENTIONS:
Device: soft peripheral defocus contact lenses — Multifocal soft contact lenses with peripheral defocus design have shown promise in reducing axial elongation. They work by reducing peripheral hyperopic defocus, which is thought to drive eye growth
  Arms: combination therapy group
Drug: Atropine 0.04% — Low-concentration atropine eyedrops (atropine 0.04% and atropine 0.01% used in this trial) are the only consistently effective pharmacological treatment for myopia control
  Arms: atropine monotherapy group; combination therapy group
Drug: Atropine (0.01%) — Low-concentration atropine eyedrops (atropine 0.04% and atropine 0.01% used in this trial) are the only consistently effective pharmacological treatment for myopia control
  Arms: control group
Device: Single Vision Spectacles — Single Vision Spectacles are the most commonly used device in high myopia children, which demonstrate better pediatric compliance, eliminate infection risks, and involve lower long-term costs.
  Arms: atropine monotherapy group; control group

SUMMARY:
Peripheral contact lens in controlling myopia progression in high myopia children（PAM）is a prospective, single-center, randomized controlled trial with three parallel arms conducted at Beijing Tongren Hospital. Chinese children aged 6-12 years with high myopia (spherical equivalent ≤-6.0D) and annual progression ≥0.75D will be enrolled. Participants will be randomized 40:40:40 to: (1) combination therapy group receiving atropine 0.04% plus soft peripheral defocus contact lenses; (2) atropine monotherapy group receiving atropine 0.04% plus spectacles; or (3) control group receiving atropine 0.01% plus spectacles. The primary outcome is change in axial length and cycloplegic refraction at 24 months. Secondary outcomes include changes in pupil diameter, and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Mainland Chinese children aged 4-16 years at enrollment
* Spherical equivalent refraction ≤-6.0D in both eyes under cycloplegia
* Astigmatism ≤2.5D in both eyes
* Anisometropia ≤2.5D
* Best corrected visual acuity ≥0.1 logMAR in both eyes
* Subject-reported non-significant ocular and systemic medical history
* Ability and willingness to wear contact lenses (for intervention groups)
* Written informed consent from parents/guardians and assent from child
* Ability to attend all scheduled follow-up visits

Exclusion Criteria:

* Previous use of myopia control treatments (atropine, orthokeratology, multifocal lenses) within 3 months
* Current use of systemic medications affecting pupil size or accommodation
* Known allergies to atropine or contact lens materials
* Current use of systemic medications that may significantly affect contact lens wear, tear film production, pupil size, adaptability, or refractive status.
* Ocular diseases: strabismus, amblyopia, glaucoma, cataract, corneal disease
* Systemic diseases affecting ocular health
* History of ocular surgery or trauma
* Inability to perform study procedures
* Participation in other clinical trials within 2 months

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Axial length elongation | from baseline to 24 months
  Axial length will be measured using the IOLMaster 500 optical biometry system (Carl Zeiss Meditec, Jena, Germany). To ensure measurement reliability and minimize random error, five consecutive measurements will be obtained for each eye at each visit, with individual measurements required to have a signal-to-noise ratio ≥2.0. The mean value of these five measurements will be calculated and used for analysis. Measurements will be standardized by time of day, conducted between 1:00 PM and 5:00 PM at all visits to minimize the influence of diurnal variations in axial length.

SECONDARY OUTCOMES:
Change in cycloplegic spherical equivalent refraction | Baseline, 6 months, 12 months, 18 months, and 24 months.
  The change in spherical equivalent refraction (SE = sphere + cylinder/2) under cycloplegia, measured from baseline. Cycloplegia will be induced using compound tropicamide eyedrops per a standardized protocol and confirmed by pupil diameter (≥6 mm) and light reflex assessment. Refraction will then be measured using an autorefractor (Topcon KR-8800). Five measurements will be taken per eye, and the mean SE will be calculated from readings with a divergence of less than 0.25 D.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Eye Center, Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No